CLINICAL TRIAL: NCT01577706
Title: Spectroscopic Imaging of GABA and Glutamate/Glutamine in Healthy Volunteers at 4T: A Double Blind, Crossover Drug Challenge Study
Brief Title: Spectroscopic Imaging at 4T: A Drug Challenge Study
Acronym: CEBRA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, John Eric Nestler Jensen, Associate Biophysicist, Director-High Field Imaging and Spectroscopy Program, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012P000197
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: AOD Effects and Consequences
Keywords: GABA; glutamate; glutamine; spectroscopy; brain; imaging; alprazolam; dextroamphetamine; placebo
MeSH Terms: interventions — Alprazolam; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alprazolam (A) (Active Comparator): Alprazolam (Xanax), gel-capsule, 1mg, single-dose, 1-day
  Interventions: Drug: Alprazolam
- Dextroamphetamine (D) (Active Comparator): Dextroamphetamine (Dexedrine), gel-capsule, 20mg, single-dose, 1-day
  Interventions: Drug: Dextroamphetamine
- Placebo (P) (Placebo Comparator): Placebo gel-capsule, single-dose, 1-day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprazolam — Alprazolam, gel-capsule, 1mg, single-dose, 1-day
  Other Names: Xanax
  Arms: Alprazolam (A)
Drug: Dextroamphetamine — Dextroamphetamine, gel-capsule, 20mg, single-dose, 1-day
  Other Names: Dexedrine
  Arms: Dextroamphetamine (D)
Other: Placebo — Placebo, gel-capsule, single-dose, 1-day
  Arms: Placebo (P)

SUMMARY:
An advanced technique for rapid magnetic resonance proton spectroscopic imaging (1H-MRSI) will be employed in a drug challenge study in healthy volunteers to spatially map and measure acute changes in the brain chemicals GABA, glutamate and glutamine after administration of a drug. Three condition will be tested in a double-blind fashion, i)depressant, ii)stimulant, iii)placebo. It is hypothesized that unique and reproducible spatial and directional metabolic response patterns will be observed, unique to each condition within the brain.

DETAILED DESCRIPTION:
Proton magnetic resonance spectroscopy (1H MRS) is a powerful tool for assessing neurochemistry non-invasively in vivo. However, the primary shortcoming in most studies is the lack of spatial coverage afforded by the typical single-voxel design. Limits on participant tolerance and financial resources restrict single-voxel studies to an examination of one or two carefully chosen voxels per scan, thus inadequately addressing the question of focal vs. global pathophysiology. A secondary shortcoming is that most studies report on either GABA or glutamate-glutamine (Glu-Gln) due to the technically demanding spectral-editing techniques that must be implemented in order to resolve and quantify those metabolites with any accuracy.

1H MRS imaging (MRSI) can partially overcome these limitations by providing a global picture of brain chemistry rather than just the focal snapshot afforded by the single-voxel design. However, the scan time necessary for collecting enough data for adequate spatial resolution and signal-to-noise, particularly if also using specialized spectral-editing techniques, is still too lengthy. We recently developed a method that combines Spectroscopic Imaging with the MEGAPRESS-based difference-editing acquisition for optimal GABA detection as well as for optimal detection of Glu and Gln. This MEGACSI sequence will permit us to obtain the maximum amount of neurochemical information in a clinically sound scan time, while using the current state-of-the-art MRS editing methods for optimal detection of GABA, Glu, and Gln.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male volunteers between the ages of 21-45
* Non-smoking participants are preferred, but will admit those who smoke less than 5 cigarettes per day
* Participants must be able to read screening materials including consent form and give informed consent

Exclusion Criteria:

* Participants cannot meet DSM-IV criteria for lifetime and/or current mood, anxiety, psychotic, and alcohol/drug use disorders as identified by the SCID
* Participants cannot be taking any prescription medication (except oral contraceptives, certain short-term anti-fungal agents, and some topical creams for dermal conditions) or nutritional supplements
* Participants cannot be taking any psychotropic medications
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participants cannot have any conditions that are contraindicated for MRI
* Participants cannot have a family history of alcoholism
* Participants cannot have any abnormal blood chemistries/urinalysis results or any other medical condition that may affect drug disposition (e.g., Hepatitis C)
* Participants cannot have current or past cardiac problems, and they also cannot have a family history of sudden death or ventricular arrhythmia
* Participants who, in the investigators' judgment, will not likely be able to comply with the study protocol.
* Participants cannot have any clinically significant findings in the structural anatomic brain scans (per the MRI report read by a board-certified radiologist).

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Jensen, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Imaging Center, McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
At present, there is no plan to share IPD data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Dextroamphetamine, Alprazolam, Placebo Sequence; Alprazolam, Dextroamphetamine, Placebo Sequence; Placebo, Dextroamphetamine, Alprazolam Sequence: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Alprazolam: Alprazolam, gel-capsule, 1mg, single-dose, 1-day Dextroamphetamine: Dextroamphetamine, gel-capsule, 20mg, single-dose, 1-day
  Placebo: single-dose, 1-day
Period: First Intervention (1 Day)
Arm/Group | Dextroamphetamine, Alprazolam, Placebo Sequence | Alprazolam, Dextroamphetamine, Placebo Sequence | Placebo, Dextroamphetamine, Alprazolam Sequence
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0
Period: Washout (at Least 1 Week)
Arm/Group | Dextroamphetamine, Alprazolam, Placebo Sequence | Alprazolam, Dextroamphetamine, Placebo Sequence | Placebo, Dextroamphetamine, Alprazolam Sequence
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Dextroamphetamine, Alprazolam, Placebo Sequence | Alprazolam, Dextroamphetamine, Placebo Sequence | Placebo, Dextroamphetamine, Alprazolam Sequence
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0
Period: Washout (at Least 1 Week)
Arm/Group | Dextroamphetamine, Alprazolam, Placebo Sequence | Alprazolam, Dextroamphetamine, Placebo Sequence | Placebo, Dextroamphetamine, Alprazolam Sequence
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Dextroamphetamine, Alprazolam, Placebo Sequence | Alprazolam, Dextroamphetamine, Placebo Sequence | Placebo, Dextroamphetamine, Alprazolam Sequence
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
Groups:
- All Study Participants: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Alprazolam: Alprazolam, gel-capsule, 1mg, single-dose, 1-day
  Dextroamphetamine: Dextroamphetamine, gel-capsule, 20mg, single-dose, 1-day
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Left Thalamus: Percent Change in GABA Levels After an Acute Drug Challenge
Description: The primary goal of this study is to assess the efficacy of an advanced spectroscopic imaging protocol in detecting changes in the levels of brain GABA in response to an acute drug challenge.
  GABA levels are expressed as a ratio to total creatinine: GABA/Cr percent change = 100*(later timepoint - earlier timepoint) / earlier timepoint
Time Frame: from 45 minutes post-dose to 102 minutes post-dose in 19-minute intervals (4 time points at t1: 45, t2: 64, t3: 83, t4: 102 minutes post-dose)
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Placebo: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Placebo: single-dose, 1-day
- Alprazolam: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Alprazolam: Alprazolam, gel-capsule, 1mg, single-dose, 1-day
- Dextroamphetamine: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Dextroamphetamine: Dextroamphetamine, gel-capsule, 20mg, single-dose, 1-day
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min | -6.80 [-21.48 to 16.18] | 23.57 [-1.97 to 64.94] | -12.51 [-21.04 to 21.22]
  t1 to t3: 45min-83min | -2.63 [-7.82 to 16.87] | 39.29 [29.17 to 50.69] | 8.26 [-8.12 to 46.09]
  t1 to t4: 45min-102min | 10.01 [-25.15 to 25.52] | 23.30 [17.75 to 58.61] | 13.63 [-1.96 to 44.44]
  t2 to t3: 64min-83min | 4.47 [-16.73 to 52.66] | 12.72 [1.46 to 37.76] | 17.75 [5.02 to 30.20]
  t3 to t4: 83min-102min | -6.32 [-20.28 to 32.66] | -2.10 [-10.90 to 9.20] | 5.45 [-22.42 to 25.76]
  t2 to t4: 64min-102min | 15.44 [-16.72 to 47.92] | 10.79 [-4.71 to 44.32] | 24.16 [-0.26 to 38.62]

2. Primary Outcome: Left Basal-Ganglia: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min | -2.91 [-32.57 to 40.70] | 43.17 [12.28 to 47.33] | 5.28 [-6.26 to 39.08]
  t1 to t3: 45min-83min | 2.11 [-12.57 to 24.86] | 43.09 [0.95 to 121.66] | 17.06 [-8.04 to 58.61]
  t1 to t4: 45min-102min | 15.59 [-24.01 to 47.89] | 44.26 [26.85 to 57.43] | 14.68 [-24.68 to 80.77]
  t2 to t3: 64min-83min | -0.58 [-31.51 to 49.01] | 6.57 [-7.83 to 35.21] | 13.40 [-1.90 to 14.04]
  t3 to t4: 83min-102min | 2.66 [-23.72 to 99.09] | 3.53 [-30.30 to 42.90] | 20.19 [-32.47 to 47.63]
  t2 to t4: 64min-102min | 5.10 [-21.73 to 45.14] | -4.57 [-25.72 to 28.48] | 22.34 [3.56 to 32.70]

3. Primary Outcome: Left Temporal: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Population: One participant is missing GABA level at t4 while on Placebo, and one participant is missing GABA level at t2 while on Alprazolam.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min: number analyzed (Participants) | 7 | 6 | 7
  t1 to t2: 45min-64min | -10.24 [-30.56 to 97.99] | 4.38 [-22.54 to 60.19] | 6.36 [-9.12 to 58.23]
  t1 to t3: 45min-83min | -13.82 [-61.55 to -10.61] | 13.44 [-18.74 to 56.65] | 1.34 [-12.22 to 15.03]
  t1 to t4: 45min-102min: number analyzed (Participants) | 6 | 7 | 7
  t1 to t4: 45min-102min | -8.77 [-17.82 to 7.78] | 58.49 [-56.01 to 98.58] | 18.24 [-15.13 to 31.52]
  t2 to t3: 64min-83min: number analyzed (Participants) | 7 | 6 | 7
  t2 to t3: 64min-83min | -10.55 [-34.46 to 24.10] | 14.55 [-2.21 to 48.14] | -6.70 [-27.30 to 15.62]
  t3 to t4: 83min-102min: number analyzed (Participants) | 6 | 7 | 7
  t3 to t4: 83min-102min | 3.83 [-4.64 to 55.05] | 32.81 [-45.86 to 44.54] | 7.53 [-20.13 to 29.78]
  t2 to t4: 64min-102min: number analyzed (Participants) | 6 | 6 | 7
  t2 to t4: 64min-102min | -2.03 [-40.16 to 1.63] | 19.68 [-43.21 to 54.55] | -20.20 [-26.64 to 15.38]

4. Primary Outcome: Parieto-Occipital: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min | 6.09 [-14.53 to 23.67] | -0.51 [-26.89 to 22.96] | 39.69 [-12.79 to 47.24]
  t1 to t3: 45min-83min | -1.60 [-13.79 to 21.08] | 1.90 [-4.50 to 13.63] | -10.29 [-21.14 to 21.33]
  t1 to t4: 45min-102min | 24.54 [-1.31 to 59.63] | 21.95 [5.90 to 41.00] | 22.35 [1.00 to 56.99]
  t2 to t3: 64min-83min | 2.15 [-20.41 to 30.46] | 4.64 [-7.82 to 37.25] | -17.33 [-41.00 to 2.01]
  t3 to t4: 83min-102min | 21.76 [15.07 to 33.23] | 10.78 [-8.66 to 33.39] | 36.38 [19.58 to 65.32]
  t2 to t4: 64min-102min | 33.46 [3.73 to 50.47] | 18.83 [3.59 to 41.72] | 7.97 [-19.53 to 26.83]

5. Primary Outcome: Right Thalamus: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Population: One participant ismissing GABA level at t4 while on Dextroamphetamine
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min | 6.55 [-6.15 to 44.75] | 2.72 [-9.20 to 8.24] | -3.61 [-28.40 to 20.53]
  t1 to t3: 45min-83min | 7.26 [3.35 to 19.28] | 19.20 [0.03 to 26.12] | 14.63 [-15.89 to 33.19]
  t1 to t4: 45min-102min: number analyzed (Participants) | 7 | 7 | 6
  t1 to t4: 45min-102min | 8.39 [-14.79 to 56.45] | 4.54 [-9.90 to 25.80] | 30.23 [20.15 to 43.23]
  t2 to t3: 64min-83min | -7.13 [-16.64 to 10.54] | 16.51 [7.97 to 35.51] | 14.95 [-13.80 to 33.15]
  t3 to t4: 83min-102min: number analyzed (Participants) | 7 | 7 | 6
  t3 to t4: 83min-102min | 2.87 [-17.56 to 31.88] | -1.78 [-24.21 to 1.69] | 1.60 [-15.84 to 4.82]
  t2 to t4: 64min-102min: number analyzed (Participants) | 7 | 7 | 6
  t2 to t4: 64min-102min | 12.69 [-9.21 to 13.71] | 12.12 [-11.69 to 38.55] | 15.51 [10.05 to 24.66]

6. Primary Outcome: Right Basal-Ganglia: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Population: One participant is missing GABA level at t4 while on Dextroamphetamine.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min | 18.63 [-13.56 to 32.90] | -9.44 [-33.69 to -1.73] | 38.78 [-20.68 to 69.65]
  t1 to t3: 45min-83min | -3.97 [-27.05 to 21.12] | 3.03 [-19.95 to 34.72] | 67.41 [4.27 to 106.38]
  t1 to t4: 45min-102min: number analyzed (Participants) | 7 | 7 | 6
  t1 to t4: 45min-102min | -1.53 [-18.69 to 146.90] | 33.58 [-7.07 to 35.39] | 37.92 [-34.20 to 69.05]
  t2 to t3: 64min-83min | -9.88 [-23.90 to 1.50] | 17.08 [4.36 to 37.09] | 21.02 [-23.89 to 43.86]
  t3 to t4: 83min-102min: number analyzed (Participants) | 7 | 7 | 6
  t3 to t4: 83min-102min | 11.46 [-18.70 to 178.53] | -0.82 [-9.81 to 37.07] | -5.96 [-20.03 to 1.13]
  t2 to t4: 64min-102min: number analyzed (Participants) | 7 | 7 | 6
  t2 to t4: 64min-102min | 10.15 [-7.73 to 64.39] | 35.96 [5.21 to 47.50] | 14.20 [-3.22 to 37.44]

7. Primary Outcome: Right Temporal: Percent Change in GABA Levels After an Acute Drug Challenge
Description: as for outcome 1
Time Frame: as for outcome 1
Population: One participant is missing GABA level at t4 while on Dextroamphetamine. Another participant is missing GABA levels both at t2 and t4 while on Dextroamphetamine. Another participant is missing GABA levels at both t2 and t4 while on Alprazolam.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alprazolam | Dextroamphetamine
Number analyzed (Participants) | 7 | 7 | 7
percent change
  t1 to t2: 45min-64min: number analyzed (Participants) | 7 | 6 | 6
  t1 to t2: 45min-64min | 14.93 [-18.14 to 48.46] | -1.45 [-19.95 to 4.29] | 2.09 [-44.68 to 40.24]
  t1 to t3: 45min-83min | 21.26 [-29.56 to 62.94] | 24.29 [-57.06 to 49.03] | -23.17 [-92.17 to 39.24]
  t1 to t4: 45min-102min: number analyzed (Participants) | 7 | 6 | 5
  t1 to t4: 45min-102min | 48.95 [5.69 to 91.43] | 31.06 [-10.94 to 62.58] | 30.23 [-48.74 to 88.02]
  t2 to t3: 64min-83min: number analyzed (Participants) | 7 | 6 | 6
  t2 to t3: 64min-83min | -13.91 [-39.87 to 21.80] | -4.86 [-16.41 to 22.82] | 18.52 [-9.25 to 42.07]
  t3 to t4: 83min-102min: number analyzed (Participants) | 7 | 6 | 5
  t3 to t4: 83min-102min | 10.85 [2.85 to 50.03] | 23.34 [9.10 to 44.14] | 70.88 [9.16 to 81.35]
  t2 to t4: 64min-102min: number analyzed (Participants) | 7 | 6 | 5
  t2 to t4: 64min-102min | 26.78 [-31.32 to 66.56] | 19.53 [2.75 to 52.00] | 31.58 [-7.14 to 122.10]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the entire clinical study which (including a no-cost extension) was of 1 year, 6 month duration, until the study closed to recruitment.
Groups:
- Placebo: Healthy male volunteers receiving drug and undergoing 1H-MRSI scanning
  Placebo, single-dose, 1-day
Arm/Group | Alprazolam | Dextroamphetamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No